CLINICAL TRIAL: NCT01225614
Title: Study of Efficacy and Tolerance of Early Launching of Nocturnal Non Invasive Ventilation in Adults With Myotonic Dystrophy Type 1(DM1)
Brief Title: Efficacy and Tolerance of Early Launching of Nocturnal Non Invasive
Acronym: DYVINE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081221; 2009-A01023-54 (IDRCB) (Other: AFSSAPS)
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Myopathy; Muscular Weakness; Respiratory Insufficiency
Keywords: Home ventilation; Myotonic dystrophy type 1 (DM1)
MeSH Terms: conditions — Muscular Diseases; Muscle Weakness; Respiratory Insufficiency; Myotonic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bipap ventilation (Experimental)
  Interventions: Device: Bilevel pressure ventilator
- Standard care (Active Comparator): Standard care and ventilation if occurrence of absolute criteria of ventilation (cf infra).
  Interventions: Device: Bilevel pressure ventilator

INTERVENTIONS:
Device: Bilevel pressure ventilator — Nocturnal home ventilation

SUMMARY:
This is a multicenter randomized controlled open labeled study testing efficacy and tolerance of early launching of night non invasive ventilation in patients with myotonic dystrophy type 1(DM1). The object of this project is to estimate the effects of the early introduction of non invasive ventilation on the arisen of complication (non expected hospitalization, tracheostomy even death) with regard to a simple respiratory follow-up in patients affected by myotonic dystrophy.

DETAILED DESCRIPTION:
DM1 is the most frequent genetic myopathy in the adult. Actually there is no curative treatment, and symptomatic cares are essentials. The respiratory impairment is the main cause of morbid-mortality at these patients. The median of survival of the patients affected by DM1 with respiratory failure is of 59 years. Mechanisms of disease are complex implying a central and a direct impairment of respiratory muscles. These patients can present an alveolar hypoventilation, notably during night, not correlated to the muscular weakness. These patients often present a cognitive impairment complicating the interpretation of the clinical symptoms and their compliance to treatments. International recommendations for launching mechanical ventilation in neuromuscular diseases are the presence: 1) at least a clinical sign of alveolar hypoventilation, and one of the following criteria 2) diurnal hypercapnia (> 45 mmHg), 3) restrictive syndrome (vital capacity < 50 % and\or maximal inspiratory pressure < 60 cmH20), 4) the existence of a oxygen night-desaturation (SaO2 < 88 %) of more than 5 minutes. However, a Cochrane meta analyzes underline the absence of randomised study estimating the profit risk in the long term of the night-mechanical ventilation for progressive myopathies such as the DM1. The validity of these criteria and the effect of the ventilation on the survival and the complications were never estimated in DM1. On a retrospective series, the compliance is inferior and the observance is only 20 % a year and the incidence of the complications (death or resort to a tracheostomy) was 6 times as important in non observant patients.

Objective (s) of the clinical study To estimate the efficiency and the tolerance of long term night-non invasive mechanical ventilation in patients affected by DM1.

Main judgment criteria:

Mortality and non programmed hospitalization.

Experimental plan:

Multicenter, national, randomized, controlled, study on 2 parallel groups. The subjects presenting a theoretical indication following consensual criteria of ventilation will be randomized either for a start up of ventilation or for an annual monitoring.

Hypothesis: Early starting of non invasive ventilation allows a reduction of 20 % of the mortality or the number of non-programmed hospitalization compared to the control group for which the rate would be 40 %.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman of age ≥ 18 years
* Preliminary medical examination
* Enlightened and written consent
* Genetically proved Steinert disease

  1. Presenting at least one of the following 3 criteria

     * A hypercapnia: PaCO2 > 45 mmHg or
     * A night-desaturation: SaO2 < 88 % more than consecutive 5 minutes or
     * Apnea syndrome with significant sleep:index of apnea / hypopnea> a 30 / hour
  2. And with presence of at least a clinical sign: dyspnoea, orthopnea, headaches, asthenia, diurnal sleepiness, or any other sign suggestive of disturbance of the sleep or of respiratory dysfunction

Exclusion Criteria:

* Age inferior to 18
* Regime of legal protection
* Pregnancy
* Absolute indication for ventilation: clinical signs (dyspnoea, orthopnea, headaches, asthenia, diurnal sleepiness), AND PaCO2 > 60 mmHg, AND night-desaturation < 88 % AND one CV < 50 % of the theoretical or the PIMAX < 60 cm H2O
* Acute respiratory failure
* Already ventilated patient
* Patient under oxygen
* Not (beneficiary to a regime of Social Security or legal successor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients having a complication (number of non expected hospitalization or death) at 5 years. | 5 YEARS
  Rate of patients having a complication (number of non expected hospitalization or death) at 5 years.

SECONDARY OUTCOMES:
Distribution of survival between the randomisation at 5 years | 5 YEARS
  Distribution of survival between the randomisation at 5 years
Number of patients having a formal indication of ventilation | 5 YEARS
  Number of patients having a formal indication of ventilation
Number of tracheostomized patients at 5 years | 5 YEARS
  Number of tracheostomized patients at 5 years
Number of non expected hospitalizations at 5 years | 5 YEARS
  Number of non expected hospitalizations at 5 years
Observance of the ventilation defined by an average minimal use of 4 am by 12:00 pm . | 5 YEARS
  Observance of the ventilation defined by an average minimal use of 4 am by 12:00 pm (determined in a objective way by the counter of the device).
Degree of respiratory and sleep impairment at 5 years | 5 YEARS
  Degree of respiratory and sleep impairment at 5 years
Quality of life SF36, scales of depression | 5 YEARS
  Quality of life SF36, scales of depression

CONTACTS AND LOCATIONS:
Overall Officials: DAVID ORLIKOWSKI, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Home ventilation unit and intensive care, centre of neuromuscular disease (Garches Mondor Necker Hendaye), Raymond Poincaré hospital Versailles Saint Quentin University., Garches, France